CLINICAL TRIAL: NCT04621604
Title: Evaluation of the Relationship Between Anti-PD-1 Exposure and Tumour VOLUME in Patients Treated for Classical HODgkin's Lymphoma.
Acronym: REVOLUMHOD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of eligible patients
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_9804_REVOLUMHOD
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Extra blood samples will be collected during chemotherapy administration to analyze pharmacokinetics of the iPD1

SUMMARY:
Anti-PD-1antibodies (iPD-1) are indicated as monotherapy in the treatment of adult patients with classical LH. The recommended dosage in LH is based on solid tumour experience and no dose-concentration-effect studies have been conducted.

According to the literature, therapeutic efficacy appears to be highly variable, and could be related to differences in treatment exposure.

Since Total metabolic tumor volume (TMTV) is a prognostic factor in LH and the clearance of iPD-1, and thus exposure to iPD-1, is related to clinical efficacy, we hypothesize that TMTV influences the exposure to iPD-1 and thus its therapeutic efficacy.

The aim of this study is to evaluate the relationship between TMTV and anti-PD-1 exposure in refractory or relapsed LH.

DETAILED DESCRIPTION:
Anti-PD-1antibodies (iPD-1), nivolumab (NIV) and pembrolizumab (PEM), act by blocking the interaction of the PD-1 receptor with its PDL1/PDL-2 ligands, which are overexpressed by tumour cells and their microenvironment, thus restoring an effective anti-tumour response. NIV and PEM are indicated as monotherapy in the treatment of adult patients with classical LH. They are administered as intravenous infusions on an outpatient basis. The recommended dosage for IVN or EMP in LH is based on solid tumour experience and no dose-concentration-effect studies have been conducted.

According to the literature, therapeutic efficacy appears to be highly variable, and could be related to differences in treatment exposure.

Since Total metabolic tumor volume (TMTV) is a prognostic factor in LH and the clearance of iPD-1, and thus exposure to iPD-1, is related to clinical efficacy, we hypothesize that TMTV influences the exposure to iPD-1 and thus its therapeutic efficacy.

The aim of this study is to evaluate the relationship between TMTV and anti-PD-1 exposure in refractory or relapsed LH. Highlighting such a relationship will make it possible to identify treatment algorithms according to the initial TMTV with a target plasma concentration defined according to the TMTV measurement. New therapeutic biomarkers would thus be highlighted.

This personalised medicine approach would make it possible to maximise the effect while reducing toxicity. This project is a first step in the implementation of a clinical study leading to recommendations for anti-PD-1 dose adaptation based on concentration and TMTV.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age
* Patient for whom anti-PD-1 antibody therapy (nivolumab or pembrolizumab) is given as monotherapy for relapsed or refractory classical Hodgkin's lymphoma within the scope of the WMA.
* Patient for whom a PET-CT for the evaluation of TMTV is available within 30 days prior to the first treatment without intercurrent antitumour therapy between the last PET-CT and the start of anti-PD1 treatment.
* For women of childbearing age, use of effective contraception
* Patient with free, informed and written consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Persons of full age subject to legal protection (judicial protection, guardianship, trusteeship), persons deprived of their liberty, pregnant or breastfeeding women, persons unable to give consent
* Patient with a contraindication to NIV or PEM treatment
* Patient previously treated with anti-PD1 regardless of indication
* Patient treated with anti-PD1 in combination with other anti-tumour treatment
* Patient participating in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Pearson's correlation between the initial Tumour Metabolic Total Volume and the area under the curve of iPD-1 . | 1 month
  linear relationship, using Pearson's correlation, between the initial Tumour Metabolic Total Volume and the area under the curve (AUC) of iPD-1 during the first treatment.

SECONDARY OUTCOMES:
Correlation between treatment exposure and initial TMTV for each cycle | 3 months
  Degree of correlation between AUC, peak concentration (Cmax), residual concentration (Cmin) measured at each treatment cycle of the first 3 months, and initial TMTV (tumour Metabolic Total Volume)
Correlation between treatment exposure and TMTV at 3 months for each cycle | 3 months
  Degree of correlation between AUC, peak concentration (Cmax), residual concentration (Cmin) measured at each treatment cycle of the first 3 months, and TMTV (tumour Metabolic Total Volume) at 3 months
Correlation between treatment exposure and response to treatment at 3 months | 3 months
  Degree of correlation between AUC, peak concentration (Cmax), and residual concentration (Cmin) measured at each treatment cycle in the first 3 months, and response to treatment as assessed by PET/CT at 3 months
Correlation between treatment exposure and cell free DNA at 3 months | 3 months
  Degree of correlation between AUC, peak concentration (Cmax), and residual concentration (Cmin) measured at each treatment cycle, and cfDNA quantification at 3 months.
Correlation between treatment exposure and PD-1 after 3 months | 3 months
  Degree of correlation between AUC, peak concentration (Cmax), and residual concentration (Cmin) measured at each treatment cycle of the first 3 months, and the expression of membrane (in the tumour before treatment) and soluble PD-1, PDL-1, and PDL-2 (in plasma before treatment and during the first 3 months of treatment)
Correlation between treatment exposure and tolerance after 3 months | 3 months
  Degree of correlation between anti-PD-1 AUC, Cmax or Cmin of anti-PD-1 at each treatment cycle in the first 3 months, and occurrence of immunological adverse events (irAE) within 3 months of starting treatment
Correlation between treatment exposure and progression-free survival | 1 year
  Degree of correlation between anti-PD-1 AUC, Cmax or Cmin of anti-PD-1 at each treatment cycle in the first 3 months, and progression-free survival
Correlation between treatment exposure and overall survival | 1 year
  Degree of correlation between anti-PD-1 AUC, Cmax or Cmin of anti-PD-1 at each treatment cycle in the first 3 months, and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Roch Houot, Pr, Principal Investigator — Rennes University Hospital
Locations (8):
- France (8):
  - CHU Angers, Angers
  - CHU Dijon, Dijon
  - CHU Nantes, Nantes
  - CH Orléans, Orléans
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Tours, Tours
  - CHBA Vannes, Vannes

IPD SHARING:
Plan to Share IPD: No